CLINICAL TRIAL: NCT05296850
Title: Investigation of the Immediate Effects of Kinesio Taping and Manual Release on Lower Extremity Performance in Young Adults With Pes Planus
Brief Title: Immediate Effects of Kinesio Taping and Manual Release in Young Adults With Pes Planus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Ertuğrul Demirdel, Assistant Professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-512
Record Dates: First submitted 2022-03-07; First posted 2022-03-25 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Pes Planus
Keywords: Pes planus; Kinesio Taping; Manual release; Plantar fascia
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial: Two parallel treatment groups; participants were randomly allocated to Group 1 [Manual release (MR)] and Group 2 [Kinesio taping (KT)]
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual release group (Experimental): Manual release will perform with plantar fascia and flexor hallucis longus stretching and tissue mobilization. Stretching/mobilization will applied for approximately 3 minutes.
  Interventions: Other: Manual Release
- Kinesio taping group (Experimental): Two techniques will be used in kinesio taping application; first technique is the gastrocnemius muscle inhibition technique and the plantar fascia ligament correction technique and other technique is the transverse arch ligament correction technique.
  Interventions: Other: Kinesio Taping

INTERVENTIONS:
Other: Manual Release — Individuals are placed in the prone position with their knees extended. The calcaneus is kept in eversion while maintaining talocrural dorsiflexion. As the toes are stretched in dorsiflexion, the therapist slides the big toe distally and proximally along the plantar fascia and flexor hallucis longus. Soft tissue mobilization depth will be applied according to the patient's tolerance and reactivity.
  Arms: Manual release group
Other: Kinesio Taping — In the first technique, an "I" tape will be applied on the plantar surface of the foot from the metatarsal heads to the popliteal fossa. First, the middle of the band is attached to the inferior of the calcaneus as the first anchor, then the ankle is dorsiflexed and the upper part of the band is applied with 15-25% tension until the popliteal fossa. The plantar fascia is placed in a stretched position by dorsiflexing the ankle and fingers, and the ends of the tape, which is divided into 4 parts, are applied separately to the metatarsal heads with 75-100% tension. In the second technique, the application is made with an "I" tape. The initial anchor starts from the dorsal aspect of the 5th metatarsal on the lateral aspect of the foot. Then, the tape passes to the medial side of the foot with 75-100% tension and is adhered to the medial side of the foot and ankle over the navicular. The end anchor is applied without tension.
  Arms: Kinesio taping group

SUMMARY:
Pes planus is a postural deformity seen with decreased medial longitudinal arch (MLA) height and this causes intense stress on the plantar fascia. Pes planus may affect individuals' activities of daily living, their productivity in occupational environments, and the risk of injury and performance in sports; It has also been reported that it may cause different musculoskeletal diseases such as plantar fasciitis, medial tibial stress syndrome, patellofemoral disorders and back pain in the future. Many clinical methods are used as a treatment for pes planus and most treatments involve supporting an overstretched plantar fascia and weakened MLA. The aim of the study is to investigate the immediate effects of kinesio taping and manual release on lower extremity performance in young adults with pes planus.

DETAILED DESCRIPTION:
This study is a randomized controlled trial, will be carried out on volunteer individuals with pes planus aged between 18-25, studying at Ankara Yıldırım Beyazıt University. Evaluation of parameters and inclusion criteria, kinesio taping and manual release applications will be made by the Physiotherapist. Individuals who meet the inclusion criteria, who volunteered to participate in the study and signed the consent sheet will be randomly divided into two groups, Group 1 [Manual Release (MR)] and Group 2 [Kinesio Taping (KT)]. A simple randomization method will be used with opaque sealed envelopes containing "1" or "2". Group allocation will be performed by an independent therapist, not involved in the study. All individuals will be evaluated with timed up-and-go test, heel rise test, 10-meter walking test, and functional reach test before and after the intervention. Manual release will be applied to group 1 after the evaluation and the evaluations will be repeated immediately the end of the application. Kinesio taping will be applied to group 2 after the evaluation and the evaluations will be repeated 45 minutes after the end of the application.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who volunteer to participate in the study
* Individuals with bilateral pes planus
* Individuals who have not had any ankle injury in the last 6 months

Exclusion Criteria:

* Individuals with severe visual and hearing impairment
* Individuals with congenital shortness or deformity in their lower extremities
* Individuals who have had any lower extremity surgery
* Individuals with hallux valgus, hallux rigidus, or calcaneal epine
* Individuals with any musculoskeletal problem other than pes planus and systemic, neurological problems
* Individuals with chronic ankle instability
* Individuals who have had problems walking for the last 6 months
* Individuals who have received treatment for pes planus in the last 6 months and use insoles

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2022-04-16 (Estimated); Study Completion 2022-04-16 (Estimated)

PRIMARY OUTCOMES:
Timed up and go test (TUG) | Change from baseline at immediately after one-session treatment
  The timed up and go test is used to assess functional mobility. The test involves getting up from a standard chair without armrests, walking around a cone 3 m in front of the chair, and returning to the original sitting position as quickly as possible without running. The test is started with the researcher's verbal "go" instruction and the time to complete the test is recorded. After a familiarization attempt, three recorded exercises are performed with one-minute rest intervals. The fastest of three attempts is saved.

SECONDARY OUTCOMES:
Heel rise test (HRT) | Change from baseline at immediately after one-session treatment
  The endurance of the gastro-soleus muscle complex is evaluated with the heel rise test. The number of toe-ups in one minute is determined when the knees of the subjects are in extension. The results are recorded as the number of repetitions.
10 meter walk test, walking speed | Change from baseline at immediately after one-session treatment
  Walking speed is evaluated with the 10 meter walking test. The test is performed at a comfortable walking pace on a 10 m walk, 14 m walkway for the start (2 m) and finish (2 m). Measurements are repeated 3 times and the average time is recorded in seconds.
10 meter walk test, cadence | Change from baseline at immediately after one-session treatment
  Cadence is evaluated with the 10 meter walking test. The test is performed at a comfortable walking pace on a 10 m walk, 14 m walkway for the start (2 m) and finish (2 m). During the 10-meter walk, the number of steps is recorded.
Functional reach test (FUT) | Change from baseline at immediately after one-session treatment
  Balance is assessed with the functional reach test. In the application of the test, the individual is asked to keep his feet open and close to a parallel shoulder-width wall. The individual have a measuring stick attached to the wall at shoulder level. The individual is asked to punch his hand and flex his shoulder 90 degrees without touching the wall, and bring the third metacarpal finger joint of his hand to the starting point of the measuring stick.The individual is guided to reach as far as possible without taking a step, without lifting his heels, without bending his knees, and the end point is recorded. The difference between the starting position and the ending position is measured in cm. The test is repeated three times and the average of the three measurements is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Ulusoy, PT, Principal Investigator — Ankara Yildirim Beyazıt University; Ertuğrul Demirdel, PhD, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım Beyazıt University, Institute of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Govind, S., Singh, K., Mahalingam, K. ve SREE Vamsi, G. To Compare the Effectiveness of Taping and Arch Support on the Flexible Flat Foot on a Random Population. Indian Journal of Forensic Medicine and Toxicology. 2020
- [Background] Okamura K, Fukuda K, Oki S, Ono T, Tanaka S, Kanai S. Effects of plantar intrinsic foot muscle strengthening exercise on static and dynamic foot kinematics: A pilot randomized controlled single-blind trial in individuals with pes planus. Gait Posture. 2020 Jan;75:40-45. doi: 10.1016/j.gaitpost.2019.09.030. Epub 2019 Sep 29. PMID 31590069
- [Background] Tas S, Unluer NO, Korkusuz F. Morphological and mechanical properties of plantar fascia and intrinsic foot muscles in individuals with and without flat foot. J Orthop Surg (Hong Kong). 2018 May-Aug;26(3):2309499018802482. doi: 10.1177/2309499018802482. PMID 30270752
- [Background] Angin S, Mickle KJ, Nester CJ. Contributions of foot muscles and plantar fascia morphology to foot posture. Gait Posture. 2018 Mar;61:238-242. doi: 10.1016/j.gaitpost.2018.01.022. Epub 2018 Mar 20. PMID 29413791
- [Background] Filardi V. Flatfoot and normal foot a comparative analysis of the stress shielding. J Orthop. 2018 Aug 16;15(3):820-825. doi: 10.1016/j.jor.2018.08.002. eCollection 2018 Sep. PMID 30140126
- [Background] Wang JS, Um GM, Choi JH. Immediate effects of kinematic taping on lower extremity muscle tone and stiffness in flexible flat feet. J Phys Ther Sci. 2016 Apr;28(4):1339-42. doi: 10.1589/jpts.28.1339. Epub 2016 Apr 28. PMID 27190479
- [Background] Montgomery G, McPhee J, Paasuke M, Sipila S, Maier AB, Hogrel JY, Degens H. Determinants of Performance in the Timed Up-and-Go and Six-Minute Walk Tests in Young and Old Healthy Adults. J Clin Med. 2020 May 21;9(5):1561. doi: 10.3390/jcm9051561. PMID 32455757
- [Background] Gunay S, Karaduman A, Ozturk BB. Effects of Aircast brace and elastic bandage on physical performance of athletes after ankle injuries. Acta Orthop Traumatol Turc. 2014;48(1):10-6. doi: 10.3944/AOTT.2014.2981. PMID 24643094
- [Background] Soulard J, Vaillant J, Balaguier R, Vuillerme N. Spatio-temporal gait parameters obtained from foot-worn inertial sensors are reliable in healthy adults in single- and dual-task conditions. Sci Rep. 2021 May 13;11(1):10229. doi: 10.1038/s41598-021-88794-4. PMID 33986307
- [Background] Tedla JS, Asiri F, Alshahrani MS, Sangadala DR, Gular K, Rengaramanujam K, Mukherjee D. Reference Values of Functional and Lateral Reach Test Among the Young Saudi Population: Their Psychometric Properties and Correlation with Anthropometric Parameters. Med Sci Monit. 2019 Jul 31;25:5683-5689. doi: 10.12659/MSM.916443. PMID 31365521
- [Background] Baltacı, G. Bantlama. (N. Ozunlu Pekyavas, Ed.). Ankara: Hipokrat Yayıncılık.2020; 194-195
- [Background] Cleland JA, Abbott JH, Kidd MO, Stockwell S, Cheney S, Gerrard DF, Flynn TW. Manual physical therapy and exercise versus electrophysical agents and exercise in the management of plantar heel pain: a multicenter randomized clinical trial. J Orthop Sports Phys Ther. 2009 Aug;39(8):573-85. doi: 10.2519/jospt.2009.3036. PMID 19687575